CLINICAL TRIAL: NCT01456494
Title: Teaching Use of Respiratory Inhalers (TURI)
Acronym: TURI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16900A
Record Dates: First submitted 2011-10-14; First posted 2011-10-20 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2018-05

CONDITIONS: Asthma; COPD
Keywords: Obstructive Lung Disease; COPD; Asthma; Inhaler; Metered-Dose Inhaler; Education; Hospital-based education
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teach-to-Goal (Experimental): Teach-to-goal (TTG) is a method of patient instruction that employs repeated rounds of teaching (demonstration, verbal, written instructions) and assessments (teach-back) of patient comprehension.
  Interventions: Other: Teach-to-Goal Education
- Brief Intervention (Experimental): A brief educational strategy that employs verbal and written instructions, without demonstration or repeated rounds of instruction, to teach patients how to use their inhalers.
  Interventions: Other: Brief Intervention

INTERVENTIONS:
Other: Brief Intervention — A brief educational strategy that employs verbal and written instructions, without demonstration or repeated rounds of instruction, to teach patients how to use their inhalers.
  Other Names: BI
  Arms: Brief Intervention
Other: Teach-to-Goal Education — Teach-to-goal (TTG) is a method of patient instruction that employs repeated rounds of teaching (demonstration, verbal, written instructions) and assessments (teach-back) of patient comprehension.
  Other Names: TTG
  Arms: Teach-to-Goal

SUMMARY:
The purpose of this study is to evaluate the feasibility of enrolling and randomizing patients into one of two educational interventions to teach appropriate respiratory inhaler technique and to collect preliminary estimates of the comparative effectiveness of two types of education.

Teach-to-Goal (TTG) education employs instruction followed by patient "teach-back," then repeated cycles of learning and assessment until a skill, i.e. respiratory inhaler technique, is mastered. By contrast, Brief Intervention (BI) education only consists of providing the patient with verbal and written instruction on the skill, i.e., respiratory inhaler technique.

The investigators hypothesize that hospital-based TTG compared to BI increases a patient's ability to learn respiratory inhaler technique. The investigators will test this hypothesis separately for the MDI and Diskus® devices.

DETAILED DESCRIPTION:
Respiratory inhalers are often used incorrectly by hospitalized patients with asthma or chronic obstructive pulmonary disease (COPD). As the mainstay of bronchodilator and anti-inflammatory therapy for these patients, the implication of this difficulty with self-management is that patients are at risk for under-treatment and worse health outcomes. Several factors are thought to contribute to poor self-management skills, particularly inadequate patient education at healthcare encounters and inadequate patient health literacy (HL; ability to understand and use healthcare instructions). Inadequate HL in patients with asthma leads to worse knowledge about medications in general and inhaler technique specifically, and patients with inadequate HL are more likely to be hospitalized. As a result, national and international guidelines for both asthma and COPD recommend patient education to improve self-management skills regarding use of respiratory inhalers and assessing patient comprehension at all points of care, including hospitals. However, the most effective strategy to instruct patients about respiratory inhaler use in hospital settings is unclear, particularly in populations enriched with inadequate HL.

Teach-to-goal (TTG) is a method of patient instruction that employs repeated rounds of teaching and assessments of patient comprehension until mastery is confirmed. Our preliminary data in hospitalized patients suggest that TTG may be a particularly powerful method to teach this high-risk population how to use respiratory inhalers correctly, including patients with inadequate HL. However, TTG is likely to be more resource-intensive (personnel training and time) than approaches used in everyday clinical settings (usual care). Further, the relative magnitude of the effectiveness of TTG compared to other less resource-intensive methods on patient comprehension and health outcomes is not known. As healthcare resources are limited, empiric data about the comparative effectiveness of TTG and alternate approaches of patient education are needed.

Therefore this pilot comparative effectiveness study will compare the TTG approach versus a brief intervention (BI) for patients hospitalized with asthma or COPD to evaluate the feasibility of conducting a randomized clinical trial of two educational interventions in this population and to collect preliminary estimates of the relative benefits of TTG vs. BI. These data will help inform the design of subsequent larger studies of comparative effectiveness.

The primary research goal is to evaluate the feasibility of conducting a randomized clinical trial of two different strategies to teach respiratory inhaler use and to determine preliminary estimates of effect size for the interventions; specifically, the investigators will assess our recruitment and retention rates, pilot test case reports and other study procedures and to evaluate the resources (staff & investigator time, costs for patient incentives and other study materials) needed to perform the trial. These data will inform subsequent studies by providing important information regarding feasibility, effect size for sample calculations and preliminary data to secure funding for the development of further research. The Specific Aims are:

Specific Aim 1: To evaluate the feasibility of enrolling and randomizing patients into an educational intervention to teach appropriate respiratory inhaler technique.

Specific Aim 2: To obtain a preliminary estimate of the effect size of TTG vs. BI in order to determine the necessary sample size for a larger comparative effectiveness study designed to improve health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Admission to the inpatient medical service and surgical service
* Physician-diagnosed asthma or COPD
* Physician plans to discharge patients home on a metered dose inhaler (MDI; e.g., albuterol)

Exclusion Criteria:

* Currently in an intensive care unit
* Physician declines to provide consent
* Patient unable to provide assent (history of cognitive impairment, unable to understand English), or declines to provide consent
* Previous participant in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie G Press, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Teach-to-Goal: Teach-to-goal (TTG) is a method of patient instruction that employs repeated rounds of teaching (demonstration, verbal, written instructions) and assessments (teach-back) of patient comprehension.
  Teach-to-Goal Education: Teach-to-goal (TTG) is a method of patient instruction that employs repeated rounds of teaching (demonstration, verbal, written instructions) and assessments (teach-back) of patient comprehension.
  N=24
- Brief Intervention: A brief educational strategy that employs verbal and written instructions, without demonstration or repeated rounds of instruction, to teach patients how to use their inhalers.
  Brief Intervention: A brief educational strategy that employs verbal and written instructions, without demonstration or repeated rounds of instruction, to teach patients how to use their inhalers.
  N=26
Period: Initial Inpatient Visit
Arm/Group | Teach-to-Goal | Brief Intervention
Started | 24 | 26
Completed | 24 | 26
Not Completed | 0 | 0
Period: Follow-Up Visit (Post 30-day Discharge)
Arm/Group | Teach-to-Goal | Brief Intervention
Started | 24 | 26
Completed | 19 | 20
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teach-to-Goal | Brief Intervention | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 22 | 37
  >=65 years | 9 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (19.0) | 51.0 (13.6) | 53.8 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 26 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 21 | 37
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Misusing Metered-Dose Inhaler (MDI) Post Education Between Teach to Goal (TTG) and Brief Intervention (BI)
Time Frame: 1 hour at the V0-V1 initial hospital study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Teach-to-Goal | Brief Intervention
Number analyzed (Participants) | 24 | 26
Participants | 3 | 12

2. Secondary Outcome: Number of Participants Misusing Diskus Post Education Between TTG and BI
Time Frame: 1 hour at the V0-V1 initial hospital study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Teach-to-Goal | Brief Intervention
Number analyzed (Participants) | 8 | 10
Participants | 2 | 8

3. Secondary Outcome: Number of Participants Reporting Acute Health-related Events 30 Days Post Hospital Discharge Between TTG and BI
Time Frame: 30 days (Visits V0-V2, ie from initial hospital visit to the 30 day post discharge phone interview)
Measure: Count of Participants; unit: Participants
Arm/Group | Teach-to-Goal | Brief Intervention
Number analyzed (Participants) | 19 | 20
Participants | 1 | 8

4. Secondary Outcome: Differences in the Prevalence of Reported Acute Health-related Events 90 Days Post Hospital Discharge Between TTG and BI
Time Frame: 90 days (from Visits V0-V3, ie from initial hospital visit to 90 days day post discharge phone interview)
Population: Due to lost to follow-up, the investigators did not collect and analyze acute health related events 90 days post discharge.
Arm/Group | Teach-to-Goal | Brief Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Self-reported Confidence With Inhaler Technique Versus Actual Technique
Description: For all patients, the investigators compared their baseline self-reported confidence using a 5-point Likert scale and whether they used their inhaler correctly. The investigators define having strong confidence as either "Agree" or "Strongly Agree" when responding to "I know how to use my inhaler correctly." The investigators define correct technique as performing 10 out of 12 steps in the inhaler technique checklist. The following statistic for each arm is for the participants who reported being confident in their inhaler technique, the number of that sub-population that demonstrated satisfactory inhaler technique
Time Frame: 1 hour at Visits V0-V1 initial hospital study visit
Population: For the TTG arm, 18 out of 24 individuals self-reported being confident in their inhaler technique. In the BI arm, 18 out of 26 reported being confident in their inhaler technique.
Measure: Count of Participants; unit: Participants
Arm/Group | Teach-to-Goal | Brief Intervention
Number analyzed (Participants) | 18 | 18
Participants | 6 | 5

ADVERSE EVENTS:
Arm/Group | Teach-to-Goal | Brief Intervention
All-Cause Mortality (participants affected / at risk) | 0/24 | 3/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes